CLINICAL TRIAL: NCT05984017
Title: A Non-interventional Study and Its Clinical Relevance With Advanced Lung Squamous Cell Carcinoma
Brief Title: A Non-interventional Study With Advanced Lung Squamous Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Deputy Director of Thoracic Oncology Department, Hunan Province Tumor Hospital
Other Study IDs: SHR-1701 RWS
Record Dates: First submitted 2023-07-31; First posted 2023-08-09 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Advanced Lung Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — needle biopsy for samples with DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No treatment is included in this study — No drug intervention or tissue sampling will be included in this study.

SUMMARY:
This is a descriptive observational study, in which data are collected in an epidemiological fashion and prospective. This study does not intend to intervene the current medical practice of the recruited patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥18 years.
* Provision of fully informed consent prior to any study specific procedures.
* Advanced or metastatic lung squamous cell carcinoma confirmed by histology or cytology.
* According to the RECIST 1.1 standard, the patient must have at least one measurable lesion.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: advanced or metastatic (stage IV) lung squamous cell carcinoma
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 2 years
  From registration onto that step until death, or censored at the date of last contact.
Overall survival | 2 years
  From registration onto that step until death, or censored at the date of last contact.

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Yongchang Zhang, Changsha, Hunan, China